CLINICAL TRIAL: NCT05217992
Title: Are There Differences Between Carriers of Haemophilia A and B? A Comparative Study of Clotting Factor Deficiencies, Bleeding Phenotype and Haemostatic Treatment Requirements
Brief Title: Are There Differences Between Carriers of Haemophilia A and B?
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/29MAR/153
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Hemophilia
Keywords: hemophilia A; hemophilia B; genetic testing; carriers
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genetic testing for hemophilia
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carriers or potential carriers of hemophilia A and B: All obligate and potential carriers among families of patient with hemophilia followed at the hemophilia treatment center of the Cliniques universitaires Saint-Luc, Brussels. Belgium
  Interventions: Other: Genetic assessment (hemophilia testing)

INTERVENTIONS:
Other: Genetic assessment (hemophilia testing) — Determination of carrier ship of hemophilia with molecular tests

SUMMARY:
This study aims to develop a systematic genetic screening strategy for (potential) female carriers of haemophilia by identifying as many female carriers as possible within the families of haemophilia patients regularly followed at Cliniques universitaires Saint-Luc (CUSL) and to search for differences between female carriers of haemophilia A (HA) and B (HB).

DETAILED DESCRIPTION:
In order to complete our local registry of female carriers, the family trees of haemophilia patients will be systematically updated during their follow-up consultations at the haemophilia centre. Female carriers not yet known in our centre, identified by the updating of pedigrees, will be invited to present themselves in the haematology consultation and to participate in the study by means of an invitation and information letter which will be given/sent to them by the index haemophilia patient. Female carriers already known for whom missing data and/or the indication of regular follow-up have been identified during the file review will also be invited to attend a consultation within the framework of the study.

At these consultations, (potential) carriers will be given information about haemophilia, the mode of genetic transmission and the implications of carrier status on patients' lives (bleeding prevention, reproductive choices, current haemophilia treatments and future prospects). We will then determine the bleeding phenotype of each patient by taking a comprehensive bleeding history. With the consent of the participants concerned, the familial genetic variant responsible for haemophilia will be sought in them in order to definitively establish their carrier status. The basal level of coagulation factors VIII (HA)/IX (HB) will also be determined. If a deficiency is found, haemostatic treatment adapted to the patient's situation will be initiated and clinical follow-up outside the study recommended.

After completion of the data collection, the data will be analyzed and compared between HA and HB carriers in order to identify possible differences between these two populations.

ELIGIBILITY:
Inclusion Criteria:

- Family member affected by haemophilia A or B and potential/obligate carriership of HA/HB.

Exclusion Criteria:

* None.

Ages: 12 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Carriers of HA/HB already known and registered at the HTC (i.e. with an EMR).
  2. Carriers identified by pedigree review, invited/informed by family related haemophilia patients registered in the HTC, accepting to participate after informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Number of carriers, bleeding phenotype in hemophilia A and B carriers | 18 month
  Comparison of bleeding phenotype between hemophilia A and B carriers, number of carriers per family confirmed at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Cedric Hermans, MD,PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, International, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krumb E, Lambert C, Van Damme A, Hermans C. Proactive systematic hemophilia carrier screening: a step toward gender equity in hemophilia care. Blood Adv. 2024 Oct 22;8(20):5268-5278. doi: 10.1182/bloodadvances.2024013866. PMID 39167764